CLINICAL TRIAL: NCT01123785
Title: A Phase I/II Multi-Center, Randomized, Double-Masked, Placebo-Controlled, Dose-Escalation Study to Evaluate the Tolerability, Safety, Pharmacokinetics, and Pharmacodynamics (Efficacy) of Chronic Twice-Daily Topical Monocular Application of INO-8875 Ophthalmic Formulation in Adults With Ocular Hypertension or Primary Open-Angle Glaucoma
Brief Title: A Dose-Escalation Study Designed to Evaluate the Tolerability, Safety, Pharmacokinetics (PK), and Efficacy of Chronic Topical Ocular Application of INO-8875 in Adults With Ocular Hypertension or Primary Open-Angle Glaucoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Inotek Pharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IPC-10-2009
Record Dates: First submitted 2010-04-27; First posted 2010-05-14 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: glaucoma; ocular hypertension; adenosine agonist; eye drop; primary open angle glaucoma
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Glaucoma, Open-Angle | interventions — INO-8875

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Matched vehicle-control
  Interventions: Drug: Placebo
- INO-8875 (Experimental): Adenosine agonist eye drop
  Interventions: Drug: INO-8875

INTERVENTIONS:
Drug: INO-8875 — eye drops for 14 days in one eye
  Arms: INO-8875
Drug: Placebo — Matched vehicle-control
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate how tolerable, safe, and effective it is to give INO-8875 eye drops to adults with glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has the diagnosis of ocular hypertension (OHT) or primary open-angle glaucoma (POAG).
2. Aged 18 to 75 years.
3. Mean intraocular pressure (IOP) of ≥24 and ≤34 mm Hg.

Exclusion Criteria:

1. No significant visual field loss or any new field loss within the past year.
2. Cup-to-disc ratio ≥0.8
3. Central corneal thickness <500 µm or >600 µm
4. History of adult asthma or chronic obstructive pulmonary disease
5. A recent (acute) or chronic medical condition that might obfuscate the Subject's study data

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2010-05; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 14 days

SECONDARY OUTCOMES:
Number of Participants with decreased Intra-ocular pressure | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Lugene Eye Institute, Glendale, California, United States